CLINICAL TRIAL: NCT07242157
Title: Effects of Topical Lidocaine and Benzocaine on Pain Level and Injection Satisfaction.
Acronym: No need
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sevil Şahin, Assoc Prof Dr, TC Erciyes University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/686
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Pain; Satisfaction; Hemodialysis; Arteriovenous Fistula
Keywords: pain; satisfaction; hemodialysis
MeSH Terms: conditions — Pain; Personal Satisfaction; Arteriovenous Fistula | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: The study population consisted of patients receiving treatment at the hemodialysis unit of a university-affiliated dialysis hospital between the study period (N = 126). Among these, 60 individuals who met the inclusion criteria and were selected using a computer-generated randomization list comprised the study sample. Sample size calculation was performed using pre-analysis data from similar studies in G*Power 3.1.9.2, assuming a 5% Type I error and 95% power, with a 39.5% difference in pain levels considered. Each study group was determined to include 18 participants
Who Masked: Participant, Investigator
Masking Description: During the data collection process, the sample of the study consisted of 60 individuals who met the inclusion criteria and were selected according to a computer-generated randomization list.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group II : Benzocain Sprey (Experimental): Benzocain Spray was applied to Experiment I group before AVF catheterization application
  Interventions: Drug: Benzocaine spray
- Group III: Placebo (Placebo Comparator): Alcohol was administered to the placebo group prior to AVF catheterization application.
  Interventions: Drug: Placebo group (control arm)
- Group 1:Lidocaine spray (Experimental): Each ml contained 10 mg lidocaine and ethanol
  Interventions: Drug: Lidocaine Spray: Each ml contained 10 mg lidocaine and ethanol. Applied to the local site to provide anesthesia

INTERVENTIONS:
Drug: Lidocaine Spray: Each ml contained 10 mg lidocaine and ethanol. Applied to the local site to provide anesthesia — In this study, a moderate, negative, and significant correlation was found between total pain scores and injection satisfaction scores in the lidocaine and benzocaine groups. Overall, evidence suggests that considering the positive effects of topical lidocaine and benzocaine on pain and satisfaction during invasive procedures represents an important step toward improving patient-centered care and satisfaction. Incorporating these interventions into clinical protocols in hemodialysis units could serve as a comfort-enhancing approach before dialysis procedures.
  Arms: Group 1:Lidocaine spray
Drug: Benzocaine spray — This study, designed to investigate the effects of lidocaine and benzocaine on reducing pain and increasing injection satisfaction during AVF catheterization, is the first of its kind conducted in Türkiye. It is expected to make a significant contribution to nursing science and provide an effective approach for nurses to reduce catheter-related pain in hemodialysis units. Nurses play a vital role in minimizing procedure-related pain, and it is essential that they possess and apply knowledge about evidence-based, easy-to-use pharmacological methods to achieve this goal.
  Arms: Group II : Benzocain Sprey
Drug: Placebo group (control arm) — Lidocaine and benzocaine sprays were provided in identical bottles with color-coded bases to maintain blinding. All participants received AVF catheterization using the same arterial and venous sites to standardize procedure-related pain. Pain (VAS) and injection satisfaction (ISS) scores were recorded immediately after the procedure.
  Arms: Group III: Placebo

SUMMARY:
This study aimed to evaluate the effectiveness of topical lidocaine and benzocaine in reducing pain and improving injection satisfaction during Arteriovenous Fistula (AVF) catheterization among hemodialysis patients.

Design:A randomized controlled trial was conducted with 60 hemodialysis patients who met the inclusion criteria.

Methods: Participants were randomly assigned into three groups: Lidocaine Spray (n=20), Benzocaine Spray (n=20), and Placebo (n=20). Pain intensity and injection satisfaction were measured immediately after catheterization using the Visual Analogue Scale (VAS) and the Injection Satisfaction Scale (ISS).

DETAILED DESCRIPTION:
All individuals included in the study were provided with private health insurance to cover any potential adverse events resulting from the procedure. The participants were informed about the study both verbally and in writing, and written informed consent forms were obtained from them. Individuals who met the inclusion criteria and signed the informed consent form were assigned to study groups according to a computer-generated randomization list based on their file numbers. Accordingly, the first group was designated as the Lidocaine Spray group (Experiment I), the second group as the Benzocaine Spray group (Experiment II), and the third group as the placebo group. The design of the study, including the formation of the groups and the implementation process, is presented in Figure 3.

Two nurses working in the hemodialysis unit volunteered to participate in the study and received training from the researcher regarding the study procedures. To eliminate individual differences, one nurse performed the Arteriovenous Fistula (AVF) catheterization, while the other collected the data. These nurses were blinded to the group assignments of the patients they intervened with. In addition, the participants themselves were unaware of the groups to which they were assigned according to computer randomization. The individuals were informed about the Visual Analog Scale and the Injection Satisfaction Evaluation Scale. The nurse responsible for data collection measured and recorded in the Case Report Form the blood pressure, pulse rate, and peripheral oxygen saturation (using a fingertip pulse oximeter) five minutes before and immediately after the procedure. Blood pressure measurements were taken from the arm opposite to the Arteriovenous Fistula (AVF) catheterization site using a calibrated digital sphygmomanometer.

Since the Lidocaine Spray and Benzocaine Spray used in the groups had similar-looking bottles, the medications were used in their original containers. For the placebo group, a Lidocaine Spray bottle was emptied, washed, and sterilized in an autoclave. The sterilized glass bottle was then filled with 70% alcohol routinely used in the hospital. Subsequently, the bottles were labeled by the researchers with color-coded bands on their bases: red for the Lidocaine Spray, blue for the Benzocaine Spray, and black for the alcohol (Figure 2). The content of each bottle was identified only by the color band on its base, known exclusively to the researchers.

To prevent errors due to catheter differences, all patients included in the study received AVF catheters. To enhance the reliability of the study and avoid variations in pain levels, the same arterial and venous catheters were used for all AVF procedures. Immediately after AVF catheterization, the patient's blood pressure, pulse rate, and peripheral oxygen saturation were measured using a fingertip pulse oximeter, and the pain intensity experienced during the procedure was recorded by the nurse on the Questionnaire Form using the Visual Analog Scale (VAS) and Injection Satisfaction Evaluation Scale (ISES) values.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years,
* non-pregnant, not planning pregnancy,
* receiving hemodialysis three times weekly for at least three months,
* continuously treated at the same institution without any change in treatment regimen,
* without pain in any part of the body affecting study outcomes,
* with a Visual Analog Scale (VAS) pain score of zero at baseline,
* no analgesics within 24 hours prior,
* a baseline Algometer pressure pain threshold of 8-16 lbs.
* participants were required to understand Turkish,
* communicate effectively,
* volunteer for the study, and
* provide written informed consent.

Exclusion Criteria:

* Individuals with neurological disorders such as epilepsy, Alzheimer's disease, Parkinson's disease, or multiple sclerosis,
* unable or unwilling to comply with study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Pain level (Visual Anolog Scale) | Evaluation was made immediately after application
  The Visual Analog Scale (VAS) is a widely used, subjective measurement tool designed to assess the intensity of pain or other symptoms that cannot be directly quantified. It typically consists of a 10-cm horizontal line with two anchor points at each end, representing the extremes of the symptom being measured-commonly "no pain" (0 cm) and "worst imaginable pain" (10 cm). Participants are asked to mark a point on the line that best reflects the severity of their current experience.
  The distance (in centimeters or millimeters) between the left anchor and the participant's mark is measured to obtain the VAS score. Higher scores indicate greater symptom intensity. The VAS is considered a reliable and valid instrument due to its simplicity, sensitivity to change, and ability to capture nuanced variations in subjective experiences. It is frequently used in clinical and research settings, particularly in pain assessment, postoperative evaluation, and intervention studies.

SECONDARY OUTCOMES:
Injection Satisfaction Scale | Evaluation was made immediately after application
  The Injection Satisfaction Scale is a standardized instrument used to evaluate an individual's level of satisfaction with injection-related procedures. The scale assesses multiple dimensions of the injection experience, including perceived comfort during the injection, ease of administration, overall acceptability, and the individual's willingness to undergo the same procedure again. It is typically administered immediately after the injection to minimize recall bias.
  Items on the scale are rated using a Likert-type response format, with higher scores indicating greater satisfaction. The scale has been shown to be a reliable and valid measure for assessing patient-reported outcomes related to injection procedures across various clinical and research settings. Its use allows for a comprehensive evaluation of patient satisfaction, facilitating comparisons between different injection techniques, devices, or interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes Universty, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37820220/